CLINICAL TRIAL: NCT00922493
Title: Weaning Process in Elderly Intubated Patients Submitted to Inspiratory Muscle Training
Brief Title: Inspiratory Muscle Training in Weaning
Acronym: IMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Euro-American Network of Human Kinetics (Other)
Allocation: Randomized | Model: Parallel
Other Study IDs: 250525
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Weaning
Keywords: weaning; inspiratory muscle training; maximum inspiratory pressure (MIP); index of Tobin (IT); intubated; intensive care unit; elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: inspiratory muscle training — Protocol of inspiratory muscle training using threshold IMT®: After the MIP was measured, inspiratory muscle training was initiated. The Threshold-IMT® device of a linear pressure load produces a resistance to inspiration through the use of a flow-independent one-way valve. During expiration there is no resistance because the unidirectional valve opens, while during inspiration the valve closes, becoming "hard" due to the resistance of the spring. The suggested protocol was: initial load of 30% of the M24, increasing daily by 10%, with training for five minutes, twice a day, seven times a week in the period from the beginning of the weaning from the MV until the extubation of the patient.
  An essential factor was the use of supplemental oxygen (O2) as needed by the patient. The patients were in DD with fowler 45º.

SUMMARY:
Background: the objective of the present inquiry was to evaluate the weaning process in intubated older people subjected to inspiratory muscle training and to correlate the predictors of ventilatory interruption with its success.

Methods: the patients were divided randomly into an experimental group (EG, n=14; age=82±4 years) that received conventional physiotherapy plus inspiratory muscle training (IMT) with threshold IMT® and a control group (CG, n=14; age=81±6 years) that received only conventional physiotherapy. The predictors evaluates were the maximum inspiratory pressure (MIP) and the index of Tobin (IT). The protocol for muscle training consisted of an initial load of 30% MIP, which was increased by 10% daily; training was administered for five minutes, twice a day, seven times a week with supplemental oxygen for the entire period from the decision to wean up to extubation.

DETAILED DESCRIPTION:
The sample for this investigation was selected in a randomized way in the period between December 2007 and November 2008. The individuals were successively entered in the research as they were admitted to the ICU, in respect of the criteria of inclusion and exclusion. From the total number of admitted patients in the period (n=67), many were excluded because they had been tracheostomized (n=25), were dead (n=13) or were transferred out of the hospital (n=1). Those that remained intubated (n=28) and went to the spontaneous mode were chosen randomly and in alternating fashion were divided into the experimental group (EG) or the control group (CG). The EG (n=14; age=82±4 years-old) underwent conventional physiotherapy plus inspiratory muscular training with threshold IMT® (Respironics/EUA - 2004), and the CG (n=14; age=81±6 years-old) received only conventional physiotherapy with no intervention that favored the inspiratory muscle strengthening.

As inclusion criteria, the individuals of the sample were required to have undergone MV for at least 48 hours in a controlled way13, as intubation is diagnostic for acute respiratory injury type 1 and has a maximum value of MIP of -20 cmH2O16.

Exclusion criteria included any type of acute condition (cardiac arrhythmia) or chronic condition, such as insufficient congestive heart failure or unstable ischemic cardiac disease17, that could compromise weaning or could impede the accomplishment of inspiratory muscle training (neuropathy and myopathy). Tracheostomized patients (in the pre-test), those with neurological problems (cerebral vascular accident, cerebrospinal trauma or spinal medullar trauma), those with morbid obesity or those taking medicine that could cause a disorder of attention, as well as cases of auto-extubation, were also excluded.

The criteria of inclusion and exclusion were evaluated via examination of the patients' medical records and physical examination daily and in each session. The daily adherence of the patients to the necessary parameters for the study was noted for each patient.

ELIGIBILITY:
Inclusion Criteria:

* the individuals of the sample were required to have undergone Mechanical Ventilation for at least 48 hours in a controlled way
* intubation is diagnostic for acute respiratory injury type 1
* has a maximum value of MIP of -20 cmH2O16

Exclusion Criteria:

* any type of acute condition (cardiac arrhythmia) or chronic condition, such as insufficient congestive heart failure or unstable ischemic cardiac disease, that could compromise weaning or could impede the accomplishment of inspiratory muscle training (neuropathy and myopathy).
* Tracheostomized patients (in the pre-test).
* patients with neurological problems (cerebral vascular accident, cerebrospinal trauma or spinal medullar trauma.
* patients with morbid obesity
* patients taking medicine that could cause a disorder of attention.
* cases of auto-extubation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-12; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the MIP

SECONDARY OUTCOMES:
Measurement of rapid shallow breathing (IT)

CONTACTS AND LOCATIONS:
Locations (1):
- Quinta D'or Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Cader SA, Vale RG, Castro JC, Bacelar SC, Biehl C, Gomes MC, Cabrer WE, Dantas EH. Inspiratory muscle training improves maximal inspiratory pressure and may assist weaning in older intubated patients: a randomised trial. J Physiother. 2010;56(3):171-7. doi: 10.1016/s1836-9553(10)70022-9. PMID 20795923